CLINICAL TRIAL: NCT04314414
Title: Peer Recovery Coaching to Facilitate Comprehensive HCV, HIV and Opioid Use Disorder Treatment: A Pilot Study
Brief Title: Coaching for HCV and HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-39712; 1UL1TR001430 (NIH); 5P30AI042853 (NIH)
Record Dates: First submitted 2020-03-13; First posted 2020-03-19 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-11

CONDITIONS: Hepatitis C; HIV Infections; Opioid-use Disorder
Keywords: Peer recovery coach (PRC); Pre-exposure prophylaxis (PrEP); HIV care; HCV care; Low-barrier-to-access (LBA)
MeSH Terms: conditions — Hepatitis C; HIV Infections; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants in the intervention group will receive a semi-scripted brief motivational interview from the peer recovery coach (PRC) in addition to the standard of care at Boston Medical Center (BMC) for HIV, HCV, and opioid use disorder.
  Interventions: Other: PRC brief motivational interview intervention; Other: Phone contact

INTERVENTIONS:
Other: PRC brief motivational interview intervention — The intervention will involve the following elements: establishing rapport, asking permission to discuss drugs, discussing the pros and cons associated with drug use, uncovering the gaps between current and desired quality of life and determining readiness to change. The intervention will last approximately 20 minutes and take place at the time of the clinical visit while participants are waiting to be seen by a clinician or are awaiting laboratory testing.
Other: Phone contact — The PRC will remain in at least weekly contact by phone with each participant.

SUMMARY:
The objective of this study is to determine the feasibility and acceptability of a peer recovery coach (PRC) intervention to improve linkage to hepatitis C (HCV) and/or human immunodeficiency virus (HIV) care, treatment initiation, and evaluation for HIV pre-exposure prophylaxis (PrEP) (when applicable) among individuals with a history of opioid use disorder accessing a substance use low-barrier-to-access (LBA) walk-in clinic.

In-depth interviews will be administered to participants at baseline, three- and six-months for study participants (40 total participants). The investigator will also follow-up with the per recovery coach and administer surveys to assess the feasibility of a peer recovery coaching intervention in improving HCV/HIV related linkage to care and management. Patient medical records and peer recovery coach monthly reports will be accessed and reviewed to determine fidelity to research protocols.

DETAILED DESCRIPTION:
*NOTE* Due to the COVID-19 pandemic, surveys were conducted via telephone and not all participants could be contacted. Therefore, the number of results from participants at three months and six months vary. The data gathered are from participants that were reachable and completed the surveys.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with opioid use disorder, non-reactive HIV antibody test and reactive HCV antibody testing at the BMC LBA walk-in clinic
* Able to speak English
* Individuals providing contact information of two family members or friends
* Individuals signing a medical records release form

Exclusion Criteria:

* Individuals already linked to substance use care
* Individuals co-infected with HIV and HCV and engaged in care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-12-20 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina A Assoumou, MD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center - Low-Barrier-Access (LBA) walk-in clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Participants in the intervention group will receive a semi-scripted brief motivational interview from the peer recovery coach (PRC) in addition to the standard of care at Boston Medical Center (BMC) for HIV, hepatitis C (HCV), and opioid use disorder.
  PRC brief motivational interview intervention: The intervention will involve the following elements: establishing rapport, asking permission to discuss drugs, discussing the pros and cons associated with drug use, uncovering the gaps between current and desired quality of life and determining readiness to change. The intervention will last approximately 20 minutes and take place at the time of the clinical visit while participants are waiting to be seen by a clinician or are awaiting laboratory testing.
  Phone contact: The PRC will remain in at least weekly contact by phone with each participant.
Period: 3 Months
Arm/Group | Intervention Group
Started | 31
Completed | 31
Not Completed | 0
Period: 6 Months
Arm/Group | Intervention Group
Started | 31
Completed | 29
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  How would you describe your racial/ethnic identity? (check all that apply): American Indian or Alaska Native | 2
  How would you describe your racial/ethnic identity? (check all that apply): Asian | 0
  How would you describe your racial/ethnic identity? (check all that apply): Black or African American | 3
  How would you describe your racial/ethnic identity? (check all that apply): Native Hawaiian or Pacific Islander | 1
  How would you describe your racial/ethnic identity? (check all that apply): Hispanic/Latinx | 8
  How would you describe your racial/ethnic identity? (check all that apply): White | 17
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention
Description: As part of an investigator developed survey a 5-point LIkert scale question will be asked on how acceptable the intervention/care was where 1 is not acceptable and 5 is very acceptable.
Time Frame: 6 months
Population: 20 out of the 29 participants that were retained at 6 months, completed the 6 month satisfaction survey. 9 Participants were unreachable at 6 months.
  Only 14 participants were asked about the cell phones as it was added later in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 29
Participants
  Satisfaction working with Peer Recovery Coach: number analyzed (Participants) | 20
  Satisfaction working with Peer Recovery Coach: Very Satisfied/Strongly Agreed | 13
  Satisfaction working with Peer Recovery Coach: Satisfied/Agreed | 6
  Satisfaction working with Peer Recovery Coach: Neither Satisfied nor Dissatisfied/NA | 0
  Satisfaction working with Peer Recovery Coach: Dissatisfied/Disagreed | 0
  Satisfaction working with Peer Recovery Coach: Very Dissatisfied/Strongly Disagreed | 1
  Intervention was helpful: number analyzed (Participants) | 20
  Intervention was helpful: Very Satisfied/Strongly Agreed | 16
  Intervention was helpful: Satisfied/Agreed | 3
  Intervention was helpful: Neither Satisfied nor Dissatisfied/NA | 1
  Intervention was helpful: Dissatisfied/Disagreed | 0
  Intervention was helpful: Very Dissatisfied/Strongly Disagreed | 0
  Peer Recovery Coach Provided Navigation to Substance Use Programs/Resources: number analyzed (Participants) | 20
  Peer Recovery Coach Provided Navigation to Substance Use Programs/Resources: Very Satisfied/Strongly Agreed | 15
  Peer Recovery Coach Provided Navigation to Substance Use Programs/Resources: Satisfied/Agreed | 4
  Peer Recovery Coach Provided Navigation to Substance Use Programs/Resources: Neither Satisfied nor Dissatisfied/NA | 0
  Peer Recovery Coach Provided Navigation to Substance Use Programs/Resources: Dissatisfied/Disagreed | 0
  Peer Recovery Coach Provided Navigation to Substance Use Programs/Resources: Very Dissatisfied/Strongly Disagreed | 1
  Peer Recovery Coach Provided Access to HIV Prevention and PrEP: number analyzed (Participants) | 20
  Peer Recovery Coach Provided Access to HIV Prevention and PrEP: Very Satisfied/Strongly Agreed | 12
  Peer Recovery Coach Provided Access to HIV Prevention and PrEP: Satisfied/Agreed | 7
  Peer Recovery Coach Provided Access to HIV Prevention and PrEP: Neither Satisfied nor Dissatisfied/NA | 1
  Peer Recovery Coach Provided Access to HIV Prevention and PrEP: Dissatisfied/Disagreed | 0
  Peer Recovery Coach Provided Access to HIV Prevention and PrEP: Very Dissatisfied/Strongly Disagreed | 0
  Helpfulness of Phone: number analyzed (Participants) | 14
  Helpfulness of Phone: Very Satisfied/Strongly Agreed | 12
  Helpfulness of Phone: Satisfied/Agreed | 2
  Helpfulness of Phone: Neither Satisfied nor Dissatisfied/NA | 0
  Helpfulness of Phone: Dissatisfied/Disagreed | 0
  Helpfulness of Phone: Very Dissatisfied/Strongly Disagreed | 0
  Lived-Experience of Peer Recovery Had Positive Impact: number analyzed (Participants) | 20
  Lived-Experience of Peer Recovery Had Positive Impact: Very Satisfied/Strongly Agreed | 15
  Lived-Experience of Peer Recovery Had Positive Impact: Satisfied/Agreed | 4
  Lived-Experience of Peer Recovery Had Positive Impact: Neither Satisfied nor Dissatisfied/NA | 0
  Lived-Experience of Peer Recovery Had Positive Impact: Dissatisfied/Disagreed | 0
  Lived-Experience of Peer Recovery Had Positive Impact: Very Dissatisfied/Strongly Disagreed | 1

2. Secondary Outcome: Participant Linkage to HIV Care
Description: Participants will be interviewed and asked investigator developed questions about linkage to HIV care
Time Frame: 3 months and 6 months
Population: At 3 months 31 participants retained in the study, but only 16 participants completed the 3 month satisfaction survey due to unable to contact all participants.
  At 6 months 29 participants retained in the study but only 20 completed the 6 month satisfaction survey due to unable to contact all participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
Participants
  3 Months: PRC provided access to HIV prevention and PrEP.: number analyzed (Participants) | 16
  3 Months: PRC provided access to HIV prevention and PrEP.: Strongly Agree | 9
  3 Months: PRC provided access to HIV prevention and PrEP.: Agree | 5
  3 Months: PRC provided access to HIV prevention and PrEP.: Neither/Na | 2
  3 Months: PRC provided access to HIV prevention and PrEP.: Disagree | 0
  3 Months: PRC provided access to HIV prevention and PrEP.: Strongly | 0
  6 Months: PRC provided access to HIV prevention and PrEP.: number analyzed (Participants) | 20
  6 Months: PRC provided access to HIV prevention and PrEP.: Strongly Agree | 12
  6 Months: PRC provided access to HIV prevention and PrEP.: Agree | 7
  6 Months: PRC provided access to HIV prevention and PrEP.: Neither/Na | 1
  6 Months: PRC provided access to HIV prevention and PrEP.: Disagree | 0
  6 Months: PRC provided access to HIV prevention and PrEP.: Strongly | 0

3. Secondary Outcome: Participant Linkage to HCV Care
Description: Participants will be interviewed and asked investigator developed questions about linkage to HCV care
Time Frame: 6 months
Population: Only 9 participants were eligible for HCV treatment as they tested positive for HCV.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
Participants
  Participants engaged in HCV treatment at time of enrollment.: number analyzed (Participants) | 9
  Participants engaged in HCV treatment at time of enrollment. | 0
  Participants receiving or had completed HCV treatment at 6 months.: number analyzed (Participants) | 9
  Participants receiving or had completed HCV treatment at 6 months. | 2

4. Secondary Outcome: Participant Linkage to Care for Opioid Use
Description: Participants will be interviewed and asked investigator developed questions about their linkage to care for opioid use
Time Frame: 3 months and 6 months
Population: At 3 months, not all participants were contactable. 16 participants out of 31 completed the satisfaction survey.
  At 6 months, not all participants were contactable. 20 participants out of 29 completed the satisfaction survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
Participants
  3 Months: The PRC provided adequate navigation to substance use programs and/or resources.: number analyzed (Participants) | 16
  3 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Strongly Agree | 10
  3 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Agree | 6
  3 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Neither or N/A | 0
  3 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Disagree | 0
  3 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Strongly Disagree | 0
  6 Months: The PRC provided adequate navigation to substance use programs and/or resources.: number analyzed (Participants) | 20
  6 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Strongly Agree | 15
  6 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Agree | 4
  6 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Neither or N/A | 0
  6 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Disagree | 1
  6 Months: The PRC provided adequate navigation to substance use programs and/or resources.: Strongly Disagree | 0

5. Secondary Outcome: Number of Participants Who Received Pre-exposure Prophylaxis (PrEP)
Description: Whether participants received PrEp treatment will be abstracted from their electronic medical records (EMR) system.
Time Frame: 6 months
Population: Of all 29 participants at 6 months, only 14 were eligible to initiate PrEP.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 29
Participants
  Number of participants that started PrEP during the intervention: number analyzed (Participants) | 14
  Number of participants that started PrEP during the intervention | 5
  Number of participants on PrEP at 6 months: number analyzed (Participants) | 14
  Number of participants on PrEP at 6 months | 6

6. Secondary Outcome: Number of Participants Who Received HCV Care
Description: Whether participants received HCV care will be abstracted from their electronic medical records (EMR) system.
Time Frame: 6 months
Population: Only 9 participants were eligible for HCV as they tested positive.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 9
Participants
  Number of participants engaged in HCV treatment at the time of enrollment | 0
  Number of participants receiving or had completed HCV treatment at 6 months. | 2

7. Secondary Outcome: Number of Participants Who Received Opioid Use Treatment
Description: Whether participants received opioid use treatment will be abstracted from their electronic medical records (EMR) system.
Time Frame: 6 months
Population: 22 participants were already on a medications for opioid use disorder (MOUD) before enrollment. Of the total number of participants analyzed, 6 started a MOUD on the day of the enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 31
Participants
  Number of participants who were on MOUD at the time of enrollment. | 22
  Number of participants that started MOUD on the day of enrollment.: number analyzed (Participants) | 9
  Number of participants that started MOUD on the day of enrollment. | 6
  Number of participants on MOUD at 6 months after enrollment | 15
  Number of participants on MOUD at enrollment and remained on through the end of the intervention: number analyzed (Participants) | 15
  Number of participants on MOUD at enrollment and remained on through the end of the intervention | 13

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT04314414/Prot_SAP_001.pdf
  • Informed Consent Form (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/14/NCT04314414/ICF_000.pdf